CLINICAL TRIAL: NCT04406428
Title: Needle-knife inciSion therApy coMpared to Usual caRe of Recurrent Esophagogastric AnastomotIc Strictures: a Multicenter Randomized Controlled Trial
Brief Title: NKI Therapy Compared to Usual Care of Recurrent Esophagogastric Anastomotic Strictures
Acronym: SAMURAI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusions
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); The Netherlands Cancer Institute (Other); Leiden University Medical Center (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL65652.091.18
Record Dates: First submitted 2020-05-25; First posted 2020-05-28 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Stricture; Anastomotic Stenosis; Dilation of Esophagus Due to Disease
MeSH Terms: conditions — Esophageal Stenosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NKI followed by EBD (Experimental)
  Interventions: Procedure: NKI followed by EBD
- Standard EBD (No Intervention)

INTERVENTIONS:
Procedure: NKI followed by EBD — Needle-knife incision therapy followed by endoscopic bougie dilation
  Arms: NKI followed by EBD

SUMMARY:
Rationale: The study hypothesizes that NKI followed by endoscopic bougie dilation therapy will result in an increased dysphagia-free period, a reduction of endoscopic procedures and dysphagia-related quality of life, and lower costs, when compared with the standard endoscopic bougie dilation (EBD) in recurrent esophagogastric anastomotic strictures.

Objective: To evaluate the efficacy and cost-effectiveness of needle-knife incision (NKI) followed by EBD compared to standard EBD in patients with recurrent esophagogastric anastomotic strictures.

Study design: This multicenter study is an randomized controlled trial in which NKI followed by EBD will be compared with standard EBD.

Study population: Patients with recurrent dysphagia (at least 1 and a maximum of 5 previous dilations) due to an anastomotic esophagogastric stricture that requires treatment with repeated endoscopic bougie dilations.

Intervention : The intervention to be investigated is the addition of NKI therapy to EBD to 18 mm esophageal diameter.

Main study parameters/endpoints: The primary outcome of this study will be EBD-free time during follow-up of 6 months. Secondary outcome parameters will be the number of endoscopic procedures for treatment of dysphagia, quality of life (QoL), cost-reduction and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent intra- or extrathoracic benign esophagogastric anastomotic stricture after esophagectomy. The definition of a stricture is based on the Ogilvie Dysphagia score (severity of dysphagia), i.e. Ogilvie score ≥2 (= ability to swallow semi-solid food or worse (Appendix table 1)).
* No patency for a standard endoscope (diameter < 10 mm)
* The recurrent stricture has been previously treated with at least 1 to a maximum of 5 EBD sessions that reached an esophageal diameter of ≥16 mm.
* The stricture should be suitable for endoscopic incision (stricture length ≤10 mm).

Exclusion Criteria:

* Benign esophageal stricture other than an esophagogastric anastomotic stricture.
* Strictures with a morphology unsuitable for NKI, such as long (>1 cm), irregulair or tortuous strictures.
* Previous endoscopic treatment of the esophageal stricture with steroid injection, incision therapy or stent placement within the past 3 months.
* Previous stent placement post-esophagectomy for anastomotic leakage.
* (Suspicion of) locally recurrent or metastasized esophageal cancer.
* Persisting postoperative esophageal fistula.
* Inability to discontinue anticoagulants or high-dose antiplatelet drugs at time of the baseline procedure. Low-dose aspirin (max. 100 mg/day) may be continued.
* Known clotting disorder that cannot pre-procedural be corrected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Dilation free time | 6 months
  EBD-free time

SECONDARY OUTCOMES:
Endoscopic procedures | 6 months
  Number of endoscopic procedures for treatment of dysphagia
QoL | 6 months
  Quality of life
Cost-reduction | 6 months
Cost-effectiveness | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No